CLINICAL TRIAL: NCT01954017
Title: A Phase Ib Randomized, Placebo Controlled Study of the Safety and Efficacy of Once Daily Dosing of STP206 in Premature Very Low Birth Weight and Extremely Low Birth Weight Neonates
Brief Title: STP206 for the Prevention of Necrotizing Enterocolitis (NEC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STP206-002
Record Dates: First submitted 2013-09-18; First posted 2013-10-01 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STP206 (Experimental): Biological
  Interventions: Biological: STP206
- Control (Placebo Comparator): Sterile water
  Interventions: Other: Control

INTERVENTIONS:
Biological: STP206 — Live Biotherapeutic
  Arms: STP206
Other: Control — Sterile Water
  Arms: Control

SUMMARY:
This study is a sequential dose escalation study to assess the safety, tolerability, and preliminary NEC-preventative efficacy of two doses of STP206 versus control in very low birth weight and extremely low birth weight neonates.

DETAILED DESCRIPTION:
Protocol STP206-002 is designed as a multi-center, randomized, double-blind, placebo controlled dose escalation study of the safety and tolerability of two doses of STP206 versus control in four sequentially decreasing birth weight strata. The primary objective of this study is to assess the safety and tolerability of once daily dosing of two dose levels of STP206 versus control in four different birth weight strata in premature neonates. Secondary objectives of this study include assessment of fecal shedding of STP206 throughout dosing and describing the incidence of NEC, incidence of relevant clinical events (sepsis/bacteremia, feeding intolerance, morbidity/complications of prematurity) and neonatal growth progression in the STP206 and control treatment groups.

Neonates for whom informed consent is obtained and who meet eligibility criteria will be eligible to enroll in this study. All neonates enrolled will receive daily doses of blinded study treatment for between 2 and 11 weeks with the duration of dosing based upon gestational age at birth. All neonates enrolled in the study will be placed under Universal Precautions and all study personnel with subject contact are trained in appropriate neonatal intensive care unit (NICU) infection control practices. While in the NICU, neonates will be evaluated daily for signs/symptoms of NEC, feeding volumes/feeding tolerance, adverse events, and concomitant medications. Physical examinations and vital signs will be performed daily during the dosing period and at the end of dosing/NICU discharge. Growth assessments will be performed every other week while in the NICU and at the end of dosing/NICU discharge. Assessments for complications of prematurity, including retinopathy of prematurity (ROP), intraventricular hemorrhage (IVH), and bronchopulmonary dysplasia (BPD) will be performed at protocol defined timeframes. Neonates enrolled in the study will have fecal/meconium samples collected daily through 4 days following the start of dosing and weekly thereafter until NICU discharge to determine fecal shedding of STP6 and STP11. Following completion of blinded study treatment dosing, neonates will be evaluated at 1 week, 4 weeks, 3 months, and 6 months for safety and growth assessments.

Neonates will be stratified into the following four birth weights: 2000-1501g, 1500 to 1000 g, 999 to 750 g and 749 to 500 g. Each birth weight stratum will contain 2 dosing groups - a low dose STP206 group and a high dose STP206 group. Within each birth weight strata/dose level, subjects will be randomized in a 2:1 ratio to the STP206 or control group. Enrollment of neonates into study groups will occur sequentially. Enrollment into the high dose group within a birth weight stratum will not proceed until after the safety data from the low dose group is reviewed by the study independent Data Safety Monitoring Committee (DSMC). Similarly, enrollment into the next lower birth weight stratum will not proceed until the safety data from the high dose group of the prior weight stratum is reviewed by the study independent Data Safety Monitoring Committee (DSMC).

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with birth weights between 2000-500g for Part A and 1500-500g for Part B
2. Ability to start treatment within four days after birth.
3. Gestational age between 23 and 32 weeks at birth
4. Obtaining of informed consent from the subject's mother after full understanding of the study purpose and procedures.
5. Parents who agree to allow the Principal Investigator and his/her staff to follow the procedures and assessments required by the protocol

Exclusion Criteria:

1. Infants with, or at high probability for, early onset sepsis (positive blood cultures or with clinical/histological chorioamnionitis with the expectation of empirical antimicrobial therapy for ≥5 days)
2. Infants with persistent pulmonary hypertension of the newborn (PPHN)
3. Congenital or chromosomal anomalies
4. Congenital or acquired gastrointestinal pathology that preclude feeds soon after birth (e.g. cleft lip is not an exclusion criterion, but a duodenal atresia is)
5. Infants in extremis to whom no further intensive care is offered by attending neonatologist (e.g., infant being provided only hospice/comfort care)
6. Other conditions of the infant which, in the opinion of the attending neonatologist, preclude participation
7. Positive maternal HIV status
8. Participation in another interventional clinical trial

   For Part A of the study, the following additional exclusion criterion will apply:
9. Small for gestational age neonates, i.e. neonates that weigh less that the 10th percentile for their gestational age according to the Estimated Fetal Weight Percentile Chart

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Caplan, MD, Principal Investigator — Endeavor Health
Locations (13):
- United States (13):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Sheridan Clinical Research / Plantation General Hospital, Sunrise, Florida
  - Augusta University, Augusta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Wesley Medical Center, Wichita, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - Medical University South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - The Medical Center of Plano, Plano, Texas
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose STP206: Biological
  STP206: Live Biotherapeutic
  ~1 billion (1 × 10^9) cfu of STP6 and ~100 million (1 × 10^8) cfu of STP11 (total of 1.1 billion cfu)
- High Dose STP206: Biological
  STP206: Live Biotherapeutic
  ~ 9 billion (9×10^9) cfu of STP6 and ~900 million (9 × 10^8) cfu of STP11 (total of 9.9 billion cfu)
Period: Overall Study
Arm/Group | Low Dose STP206 | High Dose STP206 | Control
Started | 36 | 33 | 34
Completed | 31 | 25 | 21
Not Completed | 5 | 8 | 13
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 3 | 2
Not completed — Necrotizing enterocolitis | 1 | 0 | 1
Not completed — Enteral intake stopped >7 days | 0 | 1 | 1
Not completed — All other reasons | 2 | 2 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose STP206 | High Dose STP206 | Control | Total
Number analyzed (Participants) | 36 | 33 | 34 | 103
Age, Customized [Count of Participants; unit: Participants] — Gestational Age (weeks)
  Participants
    <=28 | 24 | 16 | 23 | 63
    >28 | 12 | 16 | 10 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 14 | 38
  Male | 24 | 21 | 20 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 8 | 9 | 28
  White | 23 | 23 | 23 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
1-minute Apgar Score [Mean (Standard Deviation); unit: units on a scale] — The 1-minute Apgar score, ranging from 0 to 10, indicates how well neonates tolerate the birthing process. A higher score indicates better tolerance. Five subscales, scored from 0 to 2, are summed to obtain the total score. The neonate is assessed for activity (muscle tone), pulse, grimace, appearance (color), and respiration. Population: 1-minute Apgar scores were not obtained for all subjects.
  units on a scale
    number analyzed (Participants) | 35 | 32 | 33 | 100
    (all) | 5.1 (2.62) | 5.0 (2.04) | 4.6 (2.68) | 4.9 (2.44)
5-minute Apgar Score [Mean (Standard Deviation); unit: units on a scale] — The 5-minute Apgar score, ranging from 0 to 10, indicates how well neonates are doing 5 minutes after birth. A higher score indicates better well being. Five subscales, scored from 0 to 2, are summed to obtain the total score. The neonate is assessed for activity (muscle tone), pulse, grimace, appearance (color), and respiration. Population: 5-minute Apgar scores were not obtained for all subjects.
  units on a scale
    number analyzed (Participants) | 35 | 32 | 33 | 100
    (all) | 7.1 (1.95) | 7.5 (1.67) | 6.9 (2.18) | 7.1 (1.93)
Birth Weight [Mean (Standard Deviation); unit: grams] — Population: Birth weight data were not obtained for all subjects.
  grams
    number analyzed (Participants) | 35 | 32 | 33 | 100
    (all) | 1110.8 (422.37) | 1110.8 (408.14) | 1141.0 (434.12) | 1120.8 (415.69)

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Adverse Events Experienced by Subjects in Low-dose Treatment Groups
Description: The number and severity of adverse events, adverse events leading to study drug discontinuation, and number of deaths experienced by subjects randomized to the low-dose treatment groups
Time Frame: 30 days after the last dose of blinded study treatment
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 1a (Birth wt: 2000-1501 g) Low Dose; Group 2a (Birth wt: 1500-1000 g) Low Dose; Group 3a (Birth wt: 999-750 g) Low Dose; Group 4a (Birth wt: 749-500 g) Low Dose: Biological
  STP206: Live Biotherapeutic
  ~1 billion (1 × 10^9) cfu of STP6 and ~100 million (1 × 10^8) cfu of STP11 (total of 1.1 billion cfu)
- Group 1a (Birth wt: 2000-1501 g) Control; Group 2a (Birth wt: 1500-1000 g) Control; Group 3a (Birth wt: 999-750 g) Control; Group 4a (Birth wt: 749-500 g) Control: Sterile water
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Subjects with at least one treatment-emergent AE | 7 | 4 | 7 | 3 | 9 | 5 | 8 | 4
  Subjects with at least one treatment-related TEAE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Subjects with at least one TEAE Grade 3 | 1 | 1 | 0 | 0 | 1 | 2 | 3 | 1
  Subjects with at least one related TEAE Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects with TEAEs leading to stopping study drug | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Subjects with at least one serious adverse event | 1 | 1 | 1 | 0 | 3 | 2 | 5 | 1
  Number of deaths | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Number and Severity of Adverse Events Experienced by Subjects in High-Dose Treatment Groups
Description: as for outcome 1
Time Frame: 30 days after the last dose of blinded study treatment
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 1b (Birth wt: 2000-1501 g) High Dose; Group 2b (Birth wt: 1500-1000 g) High Dose; Group 3b (Birth wt: 999-750 g) High Dose; Group 4b (Birth wt: 749-500 g) High Dose: Biological
  STP206: Live Biotherapeutic
  ~9 billion (9 × 10^9) cfu of STP6 and ~900 million (900 × 10^8) cfu of STP11 (total of 9.9 billion cfu)
- Group 1b (Birth wt: 2000-1501 g) Control; Group 2b (Birth wt: 1500-1000 g) Control; Group 3b (Birth wt: 999-750 g) Control; Group 4b (Birth wt: 749-500 g) Control: Sterile water
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants
  Subjects with at least one treatment-emergent AE | 5 | 4 | 7 | 3 | 7 | 3 | 8 | 4
  Subjects with at least one treatment-related TEAE | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Subjects with at least one TEAE Grade 3 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 3
  Subjects with at least one related TEAE Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects with TEAEs leading to stopping study drug | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Subjects with at least one serious adverse event | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 4
  Number of deaths | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Treatment-emergent Adverse Events Experienced by Subjects in Low-Dose Treatment Groups
Description: Treatment-emergent adverse events experienced by subjects in low-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Blood: Anaemia neonatal | 1 | 0 | 2 | 1 | 5 | 2 | 2 | 0
  Blood: Anaemia | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 0
  Blood: Thrombocytopenia | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Cardiac: Foetal heart rate deceleration | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac: Bradycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cardiac: Cardio-respiratory arrest neonatal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Congenital: Ankyloglossia congenital | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Congenital: Atrial septal defect | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1
  Congenital: Patent ductus arteriosus | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Congenital: Cryptorchism | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Endocrine: Hypothyroidism | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Endocrine: Hypopituitarism | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Eye: Conjunctivitis | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Eye: Dacryostenosis acquired | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Eye: Discharge | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GI: GERD | 2 | 1 | 3 | 0 | 2 | 0 | 0 | 1
  GI: Vomiting | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0
  GI: Abdominal distension | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
  GI: Constipation | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  GI: Necrotising colitis | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GI: Diarrhoea | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  GI: Haematochezia | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  GI: Inguinal hernia | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
  GI: GI perforation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GI: Ileus | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  GI: Necrotising enterocolitis neonatal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  General: Hypothermia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  General: Generalised oedema | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  General: Infusion site extravasation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  General: Oedema | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary: Hyperbilirubinaemia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hepatobiliary: Cholestasis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Infections: Nasopharyngitis | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Infections: Pneumonia | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0
  Infections: Sepsis | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  Infections: Urinary tract infection | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Infections: Candida infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Pneumonia klebsiella | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Infections: Pneumonia staphylococcal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Acinetobacter infection | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Bacterial disease carrier | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Bacterial infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Bacterial sepsis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections: Endocarditis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Escherichia sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Neonatal pneumonia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Pneumonia escherichia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Upper respiratory tract infection | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Injury: Rib fracture | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations: Blood alkaline phosphatase incr | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations: Lab test abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations: Blood osmolarity decreased | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Investigations: Cardiac murmur | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Investigations: Haematocrit decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Investigations: Body temperature decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Investigations: Urine output decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Investigations: Blood glucose decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Investigations: Blood osmolarity increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Investigations: Chest X-ray abnormal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Investigations: Haematocrit | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Investigations: Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Metabolism: Metabolic acidosis | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1
  Metabolism: Hypoalbuminemia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Metabolism: Acidosis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Metabolism: Feeding disorder neonatal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Metabolism: Hyperphosphataemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Metabolism: Hyponatraemia | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2
  Metabolism: Hyperkalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Metabolism: Hypocalcaemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Hyperglycaemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Metabolism: Hypokalaemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Glucose tolerance impaired | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Hypernatraemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Metabolic alkalosis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Musculoskeletal: Osteopenia | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Musculoskeletal: Bone disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neoplasms: Haemangioma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Nervous system: Intraventricular haemorrhage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nervous system: Convulsion | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Perinatal conditions: Jaundice neonatal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Perinatal conditions: Neonatal disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Renal: Renal failure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Renal: Haematuria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Renal: Oliguria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Reproductive: Testicular mass | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Respiratory: Apnoea neonatal | 2 | 3 | 2 | 1 | 2 | 3 | 1 | 0
  Respiratory: Nasal congestion | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory: Apnoea | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Respiratory: Aspiration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Respiratory: Bronchopulmonary dysplasia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Respiratory: Neonatal hypoxia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Respiratory: Neonatal respiratory distress syndrom | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Respiratory: Rhinorrhoea | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory: Pulmonary haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory: Acute respiratory distress syndrome | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory: Bronchospasm | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory: Pulmonary oedema | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory: Respiratory disorder | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Skin: Dermatitis diaper | 3 | 1 | 3 | 1 | 2 | 2 | 1 | 0
  Skin: Skin discolouration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin: Skin disorder | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Skin: Blister | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Skin: Erythema | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Vascular: Venous insufficiency | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

4. Primary Outcome: Treatment-emergent Adverse Events Experienced by Subjects in High-Dose Treatment Groups
Description: Treatment-emergent adverse events experienced by subjects in high-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants
  Blood: Anaemia neonatal | 0 | 0 | 3 | 0 | 2 | 2 | 4 | 3
  Blood: Anaemia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Blood: Thrombocytopenia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Blood: Coagulopathy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Blood: Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cardiac: Foetal heart rate deceleration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cardiac: Pulmonary valve stenosis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac: Supraventricuar tachycardia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac: Tachycardia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Congenital: Patent ductus arteriosus | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Congenital: Adrenogenital syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Congenital: Laryngomalacia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Endocrine: Adrenal insufficiency | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
  Endocrine: Hypothyroidism | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Endocrine: Diabetes insipidus | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Eye: Conjunctivitis | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Eye: Retinopathy of prematurity | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Eye: Dacryostenosis acquired | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GI: GERD | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
  GI: Vomiting | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
  GI: Abdominal distension | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  GI: Constipation | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  GI: Necrotising colitis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  GI: Diarrhoea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  GI: Flatulence | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GI: Inguinal hernia | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  GI: Intestinal stenosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  GI: Umbilical hernia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  General: Hypothermia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  General: Generalised oedema | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  General: Infusion site extravasation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary: Hyperbilirubinaemia | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hepatobiliary: Cholestasis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Pneumonia | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Infections: Respiratory syncytial virus infection | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections: Sepsis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Urinary tract infection | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Infections: Candida infection | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Infections: Pneumonia klebsiella | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Pneumonia staphylococcal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Dacryocystitis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Eye infection | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Fungal sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Ophthalmia neonatorum | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Investigations: Blood osmolarity decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Investigations: Haematocrit decreased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Investigations: Blood sodium decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Investigations: Haemoglobin decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Metabolic acidosis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Metabolism: Hypoalbuminemia | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
  Metabolism: Hyponatraemia | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
  Metabolism: Hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Metabolism: Enteral feeding intolerance | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Metabolism: Hyperkalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Metabolism: Hypocalcaemia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Metabolism: Hypokalaemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Late metabolic acidosis of newborn | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Metabolism: Vitamin D deficiency | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Metabolism: Hypercalcaemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Metabolism: Hyperlipidaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Metabolism: Hypochloraemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Musculoskeletal: Osteopenia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Musculoskeletal: Bone disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neoplasms: Haemangioma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system: Intraventricular haemorrhage | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
  Nervous system: CNS ventriculitis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nervous system: Intraventricular haemorrhage neona | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nervous system: Convulsion | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Renal: Hydronephrosis | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Renal: Renal disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Renal: Renal failure acute | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Respiratory: Apnoea neonatal | 3 | 3 | 0 | 1 | 0 | 1 | 2 | 1
  Respiratory: Nasal congestion | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Respiratory: Apnoea | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory: Bronchopulmonary dysplasia | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Respiratory: Neonatal hypoxia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Respiratory: Pulmonary haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory: Apparent life threatening event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory: Pulmonary interstitial emphysema synd | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory: Stridor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Respiratory: Wheezing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Skin: Dermatitis diaper | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 0
  Skin: Rash | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin: Skin discolouration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin: Skin disorder | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Vascular: Hypotension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Grade 3 Treatment-emergent Adverse Events Experienced by Subjects in Low-Dose Treatment Groups
Description: Grade 3 treatment-emergent adverse events experienced by subjects in low-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Cardiac: cardio-respiratory arrest neonatal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Congenital: Patent ductus arteriosus | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GI: Necrotising colitis | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GI: GI perforation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections: Sepsis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Bacterial infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Bacterial sepsis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections: Endocarditis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Escherichia sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Pneumonia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Pneumonia escherichia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Respiratory: Pulmonary haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Grade 3 Treatment-emergent Adverse Events Experienced by Subjects in High-Dose Treatment Groups
Description: Grade 3 treatment-emergent adverse events experienced by subjects in high-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants
  Cardiac: Supraventricular tachycardia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GI: Necrotising colitis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  GI: Intestinal stenosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Pneumonia staphylococcal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Metabolism: Hyperkalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Renal: Renal failure acute | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Respiratory: Apparent life threatening event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

7. Primary Outcome: Serious Adverse Events Experienced by Subjects in Low-Dose Treatment Groups
Description: Serious adverse events experienced by subjects in low-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Cardiac: Cardio-respiratory arrest neonatal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Congenital: Patent ductus arteriosus | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GI: Necrotising colitis | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  GI: GI perforation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  GI: Necrotising enterocolitis neonatal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  General: Hypothermia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections: Sepsis | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Infections: Pneumonia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Bacterial infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections: Bacterial sepsis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections: Endocarditis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Escherichia sepsis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Pneumonia escherichia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections: Pneumonia klebsiella | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Nervous system: Convulsion | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Respiratory: Pulmonary haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Serious Adverse Events Experienced by Subjects in High-Dose Treatment Groups
Description: Serious adverse events experienced by subjects in high-dose treatment groups within 30 days of last exposure to study drug
Time Frame: 30 days after last administration of study drug
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants
  Cardiac: Supraventricular tachycardia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Congenital: Patent ductus arteriosus | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  GI: Necrotising colitis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Infections: Respiratory syncytial virus infection | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections: Staphylococcal sepsis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections: Pneumonia staphylococcal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system: Convulsion | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Renal: Renal failure acute | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Respiratory: Apparent life threatening event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

9. Primary Outcome: Growth Assessment Classification in Low-Dose Treatment Groups
Description: Accelerated growth area (AGA) is defined as both body weight (g) and head circumference (cm) are between 10th percentile and 90th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  Small for gestational age (SGA) SGA/Head-Spared is defined as body weight(g) is <10th percentile, and head circumference(cm) is between 10th percentile and 90th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  SGA/Head-Symmetric is defined as both body weight(g) and head circumference(cm) are <10th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  Large for gestational age (LGA) is defined as both body weight(g) and head circumference(cm) are >90th percentile according to the growth percentile charts in Appendix D of Protocol v3.0.
Time Frame: End of dosing/hospital discharge, up to 781 days
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Baseline : Number reporting | 8 | 4 | 9 | 4 | 9 | 5 | 6 | 4
  Baseline : AGA | 6 | 4 | 5 | 4 | 8 | 4 | 6 | 3
  Baseline : SGA/Head-Spared | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline : SGA/Symmetric | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline : LGA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  End of dosing/hx discharge : Number reporting | 7 | 3 | 9 | 4 | 9 | 3 | 6 | 3
  End of dosing/hx discharge : AGA | 7 | 3 | 7 | 3 | 6 | 2 | 3 | 0
  End of dosing/hx discharge : SGA/Head-Spared | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  End of dosing/hx discharge : SGA/Symmetric | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  End of dosing/hx discharge : LGA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Growth Assessment Classification in High-Dose Treatment Groups
Description: AGA is defined as both body weight (g) and head circumference (cm) are between 10th percentile and 90th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  SGA/Head-Spared is defined as body weight(g) is <10th percentile, and head circumference(cm) is between 10th percentile and 90th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  SGA/Head-Symmetric is defined as both body weight(g) and head circumference(cm) are <10th percentile according to the gender specific growth percentile charts in Appendix D of Protocol v3.0.
  LGA is defined as both body weight(g) and head circumference(cm) are >90th percentile according to the growth percentile charts in Appendix D of Protocol v3.0.
Time Frame: End of dosing/hospital discharge, up to 781 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 4
participants
  Baseline : Number reporting | 8 | 4 | 7 | 4 | 8 | 4 | 5 | 3
  Baseline : AGA | 5 | 4 | 7 | 3 | 4 | 4 | 4 | 3
  Baseline : SGA/Head-Spared | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline : SGA/Symmetric | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Baseline : LGA | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  End of dosing/hx discharge : Number reporting | 8 | 4 | 7 | 4 | 7 | 4 | 7 | 3
  End of dosing/hx discharge : AGA | 7 | 4 | 6 | 4 | 4 | 4 | 1 | 1
  End of dosing/hx discharge : SGA/Head-Spared | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  End of dosing/hx discharge : SGA/Symmetric | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
  End of dosing/hx discharge : LGA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Patients With Suspected Necrotizing Enterocolitis in Low-Dose Treatment Groups
Description: NEC is staged from I to III, from suspected to definite to advanced. The 3 stages are further divided into A (less severe) and B (more severe).
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 10 | 5 | 9 | 4
Participants
  IA | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  IB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Patients With Suspected Necrotizing Enterocolitis in High-Dose Treatment Groups
Description: as for outcome 11
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 5
Participants
  IA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  IB | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

13. Secondary Outcome: Number of Patients With Confirmed Necrotizing Enterocolitis in Low-Dose Treatment Groups
Description: as for outcome 11
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 10 | 5 | 9 | 4
Participants
  IIA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IIB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IIIA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IIIB | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Patients With Confirmed Necrotizing Enterocolitis in High-Dose Treatment Groups
Description: as for outcome 11
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 5
Participants
  IIA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IIB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IIIA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  IIIB | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

15. Secondary Outcome: Number of Patients With Sepsis in Low-Dose Treatment Groups
Description: The presence of STP6 and STP11 was assessed in peripheral blood cultures.
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants
  Present | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0
  Absent | 6 | 2 | 7 | 3 | 7 | 4 | 5 | 4
  Not evaluated | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0

16. Secondary Outcome: Number of Patients With Sepsis in High-Dose Treatment Groups
Description: The presence of STP6 and STP11 was assessed in peripheral blood cultures.
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants
  Present | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
  Absent | 8 | 4 | 7 | 4 | 6 | 4 | 5 | 4
  Not evaluated | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

17. Secondary Outcome: Number of Patients With Feeding Intolerance in Low-Dose Treatment Groups
Description: Feeding tolerance was evaluated by abdominal evaluation (any excessive distension beyond what is expected with a feed, redness of abdominal wall, firmness, presence of normal bowel sounds). Neonates placed on NPO status for at least 12 hours were considered to have feeding intolerance.
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
Participants | 2 | 1 | 2 | 0 | 6 | 2 | 8 | 2

18. Secondary Outcome: Number of Patients With Feeding Intolerance in High-Dose Treatment Groups
Description: as for outcome 17
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
Participants | 0 | 0 | 0 | 0 | 4 | 0 | 5 | 3

19. Secondary Outcome: Number of Patients With Retinopathy of Prematurity in Low-Dose Treatment Groups
Description: ROP in each eye was assessed by indirect ophthalmoscope after pupillary dilation. ROP is categorized in zones 1 to 3, the lower number representing the smallest area affected, and stages 0 to 5, the lowest number indicating the mildest form and the highest number indicating retinal detachment.
Time Frame: Start of dosing to 6 months
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 10 | 5 | 9 | 4
Participants
  Any | 0 | 0 | 1 | 1 | 7 | 3 | 5 | 4
  Zone 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Zone 2 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 3
  Zone 3 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1
  Stage 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Stage 1 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 1
  Stage 2 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2
  Stage 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Stage 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stage 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Patients With Retinopathy of Prematurity in High-Dose Treatment Groups
Description: as for outcome 19
Time Frame: Start of dosing to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 5
Participants
  Any | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 1
  Zone 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Zone 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
  Zone 3 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0
  Stage 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Stage 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Stage 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  Stage 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Stage 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stage 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Patients With Intraventricular Hemorrhage in Low-Dose Treatment Groups
Description: IVH was assessed by cranial ultrasound between the ages of 5 and 7 days and, if clinically indicated and the neonate remained hospitalized, at 28 days. IVH is graded from I to IV, with increasing severity.
Time Frame: From 5 days to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 10 | 5 | 9 | 4
Participants
  Any | 0 | 1 | 4 | 0 | 6 | 0 | 2 | 2
  Grade I | 0 | 1 | 2 | 0 | 4 | 0 | 1 | 0
  Grade II | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
  Grade III | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade IV | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

22. Secondary Outcome: Number of Patients With Intraventricular Hemorrhage in High-Dose Treatment Groups
Description: as for outcome 21
Time Frame: From 5 days to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 5
Participants
  Any | 1 | 1 | 0 | 0 | 1 | 3 | 6 | 3
  Grade I | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1
  Grade II | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1
  Grade III | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade IV | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

23. Secondary Outcome: Number of Patients With Bronchopulmonary Dysplasia in Low-Dose Treatment Groups
Description: Mild to Moderate = Need for < 30% O2 at 36 wk postmenstrual age (PMA) or discharge, whichever comes first.
  Severe = Need for ≥ 30% O2, positive pressure or both at 36 wk PMA or discharge, whichever comes first.
  For each event type, patients are counted only once if they had one or more events as this table tabulates the percentage of patients with one or more events.
Time Frame: Start of dosing to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 10 | 5 | 9 | 4
Participants
  Any | 1 | 0 | 1 | 1 | 6 | 1 | 4 | 3
  Mild to Moderate | 1 | 0 | 1 | 0 | 5 | 1 | 3 | 2
  Severe | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1

24. Secondary Outcome: Number of Patients With Bronchopulmonary Dysplasia in High-Dose Treatment Groups
Description: as for outcome 23
Time Frame: Start of dosing to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 8 | 4 | 8 | 5
Participants
  Any | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 0
  Mild to Moderate | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

25. Secondary Outcome: Number of Patients With Fecal Shedding of STP6 and STP11 in Low-Dose Treatment Groups
Description: The presence of STP6 and STP11 was assessed in fecal cultures.
Time Frame: Prior to Week 1 Day 4 and at end of dosing/hospital discharge, up to 781 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt: 2000-1501 g) Control | Group 2a (Birth wt: 1500-1000 g) Low Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3a (Birth wt: 999-750 g) Low Dose | Group 3a (Birth wt: 999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 9 | 4 | 9 | 5 | 8 | 4
participants
  Prior to Week 1 Day 4 : STP-6 | 8 | 2 | 7 | 2 | 5 | 1 | 3 | 0
  End of dosing/hx discharge : STP-6 | 6 | 2 | 6 | 0 | 6 | 0 | 3 | 0
  Prior to Week 1 Day 4 : STP-11 | 4 | 0 | 7 | 1 | 2 | 1 | 3 | 0
  End of dosing/hx discharge : STP-11 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 0

26. Secondary Outcome: Number of Patients With Fecal Shedding of STP6 and STP11 in High-Dose Treatment Groups
Description: The presence of STP6 and STP11 was assessed in fecal cultures.
Time Frame: Prior to Week 1 Day 4 and at end of dosing/hospital discharge, up to 781 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt: 2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2a (Birth wt: 1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt: 999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt: 749-500 g) Control
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 4
participants
  Prior to Week 1 Day 4 : STP-6 | 8 | 0 | 7 | 1 | 6 | 0 | 5 | 0
  End of dosing/hx discharge : STP-6 | 3 | 0 | 5 | 0 | 6 | 0 | 5 | 0
  Prior to Week 1 Day 4 : STP-11 | 8 | 0 | 7 | 0 | 5 | 0 | 5 | 0
  End of dosing/hx discharge : STP-11 | 2 | 0 | 3 | 0 | 5 | 0 | 4 | 0

ADVERSE EVENTS:
Time Frame: 6 months after last administration of study drug
Groups:
- Group 1a (Birth wt:2000-1501 g) Control; Group 2a (Birth wt:1500-1000 g) Control; Group 3a (Birth wt:999-750 g) Control; Group 4a (Birth wt:749-500 g) Control; Group 1b (Birth wt:2000-1501 g) Control; Group 2b (Birth wt:1500-1000 g) Control; Group 3b (Birth wt:999-750 g) Control; Group 4b (Birth wt:749-500 g) Control: Sterile water
- Group 2a (Birth wt:1500-1000 g) Low Dose; Group 3a (Birth wt:999-750 g) Low Dose; Group 4a (Birth wt: 749-500 g) Low Dose: Biological
  STP206: Live Biotherapeutic
  ~1 billion (1 × 10^9) cfu of STP6 and ~100 million (1 × 10^8) cfu of STP11 (total of 1.1 billion cfu)
- Group 1b (Birth wt: 2000-1501 g) High Dose; Group 2b (Birth wt: 1500-1000 g) High Dose; Group 3b (Birth wt: 999-750 g) High Dose; Group 4b (Birth wt: 749-500 g) High Dose: Biological
  STP206: Live Biotherapeutic
  ~ 9 billion (9×10^9) cfu of STP6 and ~900 million (9 × 10^8) cfu of STP11 (total of 9.9 billion cfu)
Arm/Group | Group 1a (Birth wt: 2000-1501 g) Low Dose | Group 1a (Birth wt:2000-1501 g) Control | Group 2a (Birth wt:1500-1000 g) Low Dose | Group 2a (Birth wt:1500-1000 g) Control | Group 3a (Birth wt:999-750 g) Low Dose | Group 3a (Birth wt:999-750 g) Control | Group 4a (Birth wt: 749-500 g) Low Dose | Group 4a (Birth wt:749-500 g) Control | Group 1b (Birth wt: 2000-1501 g) High Dose | Group 1b (Birth wt:2000-1501 g) Control | Group 2b (Birth wt: 1500-1000 g) High Dose | Group 2b (Birth wt:1500-1000 g) Control | Group 3b (Birth wt: 999-750 g) High Dose | Group 3b (Birth wt:999-750 g) Control | Group 4b (Birth wt: 749-500 g) High Dose | Group 4b (Birth wt:749-500 g) Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/4 | 1/9 | 0/4 | 0/9 | 0/5 | 2/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/4 | 1/8 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/4 | 2/9 | 2/4 | 3/9 | 3/5 | 5/8 | 1/4 | 1/8 | 0/4 | 2/8 | 0/4 | 2/8 | 1/4 | 4/8 | 4/4
Other Adverse Events (participants affected / at risk) | 7/8 | 4/4 | 7/9 | 3/4 | 9/9 | 5/5 | 8/8 | 4/4 | 6/8 | 4/4 | 7/8 | 3/4 | 7/8 | 3/4 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1a (Birth wt: 2000-1501 g) Low Dose (N=8) | Group 1a (Birth wt:2000-1501 g) Control (N=4) | Group 2a (Birth wt:1500-1000 g) Low Dose (N=9) | Group 2a (Birth wt:1500-1000 g) Control (N=4) | Group 3a (Birth wt:999-750 g) Low Dose (N=9) | Group 3a (Birth wt:999-750 g) Control (N=5) | Group 4a (Birth wt: 749-500 g) Low Dose (N=8) | Group 4a (Birth wt:749-500 g) Control (N=4) | Group 1b (Birth wt: 2000-1501 g) High Dose (N=8) | Group 1b (Birth wt:2000-1501 g) Control (N=4) | Group 2b (Birth wt: 1500-1000 g) High Dose (N=8) | Group 2b (Birth wt:1500-1000 g) Control (N=4) | Group 3b (Birth wt: 999-750 g) High Dose (N=8) | Group 3b (Birth wt:999-750 g) Control (N=4) | Group 4b (Birth wt: 749-500 g) High Dose (N=8) | Group 4b (Birth wt:749-500 g) Control (N=4)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Patent ductus arterioles (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1a (Birth wt: 2000-1501 g) Low Dose (N=8) | Group 1a (Birth wt:2000-1501 g) Control (N=4) | Group 2a (Birth wt:1500-1000 g) Low Dose (N=9) | Group 2a (Birth wt:1500-1000 g) Control (N=4) | Group 3a (Birth wt:999-750 g) Low Dose (N=9) | Group 3a (Birth wt:999-750 g) Control (N=5) | Group 4a (Birth wt: 749-500 g) Low Dose (N=8) | Group 4a (Birth wt:749-500 g) Control (N=4) | Group 1b (Birth wt: 2000-1501 g) High Dose (N=8) | Group 1b (Birth wt:2000-1501 g) Control (N=4) | Group 2b (Birth wt: 1500-1000 g) High Dose (N=8) | Group 2b (Birth wt:1500-1000 g) Control (N=4) | Group 3b (Birth wt: 999-750 g) High Dose (N=8) | Group 3b (Birth wt:999-750 g) Control (N=4) | Group 4b (Birth wt: 749-500 g) High Dose (N=8) | Group 4b (Birth wt:749-500 g) Control (N=4)
Anaemia neonatal (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 5 | 2 | 2 | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foetal heart rate deceleration (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Retinopathy of prematurity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Necrotising colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Milk allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acinetobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood osmolarity decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Body temperature decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood osmolarity increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Enteral feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Late metabolic acidosis of newborn (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
CNS ventriculitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Gross motor delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary dyspasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Cough (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neonatal hypoxia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT01954017/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT01954017/SAP_001.pdf